CLINICAL TRIAL: NCT02242513
Title: Ultrasound-guided Pulsed Radiofrequency Stimulation of the Tibial Nerve for Plantar Fasciitis
Brief Title: Ultrasound-guided Pulsed Radiofrequency for Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yung-Tsan Wu (Other)
Responsible Party: Sponsor-Investigator, Yung-Tsan Wu, Attending Physician, Tri-Service General Hospital
Organization: Tri-Service General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSGHIRB-2-102-05-95; TSGH-C103-115 (Other Grant/Funding Number: TSGH-C103-115)
Record Dates: First submitted 2014-09-10; First posted 2014-09-17 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Plantar Fasciitis
Keywords: Pulsed mode radiofrequency; Plantar Fasciitis; Ultrasound-guided
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Pulsed Radiofrequency Treatment; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pulsed mode radiofrequency (Active Comparator): Pulsed radiofrequency (PRF) treatment, a relative novel pain intervention at recent decade, was found to be able to alleviate pain by delivering an electrical field and heat bursts at a temperature less than 42°C to neural tissue in the absence of neural injury. One dose of PRF was given in tibial nerve behine the medial ankle in intervention group.
  Interventions: Device: Pulsed radiofrequency (PRF)
- Xylocaine (Placebo Comparator): 2 c.c xylocaine was given in tibial nerve behind the medial ankle in control group.
  Interventions: Drug: Xylocaine

INTERVENTIONS:
Device: Pulsed radiofrequency (PRF) — Pulsed radiofrequency (PRF) treatment, a relative novel pain intervention at recent decade, was found to be able to alleviate pain by delivering an electrical field and heat bursts at a temperature less than 42°C to neural tissue in the absence of neural injury.
  Other Names: Neurotherm NT1000, Neurotherm Inc., USA
  Arms: pulsed mode radiofrequency
Drug: Xylocaine
  Arms: Xylocaine

SUMMARY:
Although there are many conservative method for plantar fasciitis, patients might spend 2 years to achieve resolution. Recent study have shown that pulsed radiofrequency (PRF) lesioning of peripheral nerve can alleviate kinds of pain condition. However there are no studies of PRF lesioning of the tibial nerve in patients with plantar fascilitis by using ultrasound-guided (UG) techniques.

DETAILED DESCRIPTION:
Patients with unilateral plantar Fasciitis will be enrolled and randomized into intervention and control group. One dose of sono-guided PRF is applied in the intervention group and xylocaine in control group. Outcome measurements included visual analog scale (VAS)、foot health status questionnaire and the thickness of plantar fascile measured by musculoskeletal ultrasonography at different follow-up frame (4th week, 2nd month, 3rd month after treatment).

ELIGIBILITY:
Inclusion Criteria:

* Heel pain more than 3 months
* Age more than 20 year-old
* The increased thickness of plantar fascile (>4mm) measured by sonography
* Must be conscious
* Not receive steroid or other injection in plantar fascile in past 6 months

Exclusion Criteria:

* Cancer of any site
* Coagulopathy
* Pregnancy
* Inflammation status

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 4th, 8th and 12th weeks after treatment. | Baseline , 4th, 8th and 12th weeks after treatment.
  Using the Visual analog scale (VAS) and subscore of foot health status questionnaire to measure the pain scale before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline of functional improvement on 4th, 8th and 12th after treatment. | Baseline , 4th, 8th and 12th weeks after treatment.
  Using the functional subscore of foot health status questionnaire to measure the functional socre before treatment and multiple time frame after treatment.
Change from baseline of thickness of plantar fascile on 4th, 8th and 12th weeks after treatment. | Baseline , 4th, 8th and 12th weeks after treatment.
  Using the musculoskeletal ultrasonography to measure the thickness before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Cheng Chen, MD, MS, Study Director — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, National Defense Medical Center,
Locations (1):
- Tri-Service General Hospital, School of Medicine, National Defense Medical Center, Taipei, Neihu District, Taiwan

REFERENCES:
- [Background] Martin DC, Willis ML, Mullinax LA, Clarke NL, Homburger JA, Berger IH. Pulsed radiofrequency application in the treatment of chronic pain. Pain Pract. 2007 Mar;7(1):31-5. doi: 10.1111/j.1533-2500.2007.00107.x. PMID 17305676
- [Background] Van Zundert J, Patijn J, Kessels A, Lame I, van Suijlekom H, van Kleef M. Pulsed radiofrequency adjacent to the cervical dorsal root ganglion in chronic cervical radicular pain: a double blind sham controlled randomized clinical trial. Pain. 2007 Jan;127(1-2):173-82. doi: 10.1016/j.pain.2006.09.002. Epub 2006 Oct 18. PMID 17055165
- [Background] Rohof OJ. Radiofrequency treatment of peripheral nerves. Pain Pract. 2002 Sep;2(3):257-60. doi: 10.1046/j.1533-2500.2002.02033.x. PMID 17147740
- [Result] Thapa D, Ahuja V. Combination of diagnostic medial calcaneal nerve block followed by pulsed radiofrequency for plantar fascitis pain: A new modality. Indian J Anaesth. 2014 Mar;58(2):183-5. doi: 10.4103/0019-5049.130824. PMID 24963184
- [Result] Erken HY, Ayanoglu S, Akmaz I, Erler K, Kiral A. Prospective study of percutaneous radiofrequency nerve ablation for chronic plantar fasciitis. Foot Ankle Int. 2014 Feb;35(2):95-103. doi: 10.1177/1071100713509803. Epub 2013 Oct 28. PMID 24165571
- [Result] Sean NY, Singh I, Wai CK. Radiofrequency microtenotomy for the treatment of plantar fasciitis shows good early results. Foot Ankle Surg. 2010 Dec;16(4):174-7. doi: 10.1016/j.fas.2009.10.008. Epub 2009 Nov 25. PMID 21047605